CLINICAL TRIAL: NCT03984786
Title: Internet-delivered Cognitive Behaviour Therapy for Alcohol Misuse: A Factorial Trial Examining the Effects of Assessment Interview and Guidance
Brief Title: Internet-delivered Therapy for Alcohol Misuse: Factorial Trial of Assessment and Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Ministry of Health, Saskatchewan (Other); Saskatchewan Health Research Foundation (Other); Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-058
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Misuse
Keywords: alcohol misuse; internet; guidance; ICBT; cognitive behaviour therapy; assessment
MeSH Terms: interventions — Counseling; Ethanol

STUDY DESIGN:
Intervention Model Description: Factor 1: Guidance (yes or no)
  Factor 2: Assessment interview (yes or no)
  Each client will be randomized to one of four conditions:
  Condition 1: Assessment interview and Guidance Condition 2: Assessment Interview and No Guidance Condition 3: No Assessment Interview and Guidance Condition 4: No Assessment Interview and No Guidance
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be blinded to randomization, i.e. will not know which groups they can be randomized to. Health educators providing guidance to participants will be blinded to whether the client has been randomized to "Assessment Interview" factor (condition 1) or "No assessment interview (condition 3). All outcomes are collected online, so there is no need to blind any outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ICBT for alcohol misuse: Assessment Interview/Guidance (Experimental): In this arm, an interviewer will administer a pre-treatment assessment interview. This 30-45 minute interview will be performed after randomization during the initial telephone screen, where the interviewer will use the AUD section from SCID-5.
  Participants randomized to this arm will then receive the 8-week internet-delivered cognitive behaviour therapy (ICBT) course for alcohol misuse with guidance from a health educator through regular weekly online messages. Participants may also be contacted through emails and phone calls. The team of guides consists of registered social workers, psychologists, and graduate students, with experience delivering ICBT.
  Interventions: Behavioral: Assessment Interview; Behavioral: Guidance; Behavioral: ICBT for alcohol misuse
- ICBT for alcohol misuse: Assessment Interview/No Guidance (Experimental): In this arm, an interviewer will administer a pre-treatment assessment interview. This 30-45 minute interview will be performed after randomization during the initial telephone screen, where the interviewer will use the AUD section from SCID-5.
  Participants randomized to this arm will receive the 8-week internet-delivered cognitive behaviour therapy (ICBT) course for alcohol misuse. Participants are able to contact the Online Therapy Unit regarding any technical issues with logging onto the site. However, no guidance from a health educator will be provided. Clients will be monitored by providing brief measures on alcohol and depression each week. However, clients will only be contacted if there is a significant clinical issue requiring attention (e.g., sudden increase in symptoms of depression and suicidal ideation).
  Interventions: Behavioral: Assessment Interview; Behavioral: ICBT for alcohol misuse
- ICBT alcohol misuse: No Assessment Interview/Guidance (Experimental): The client will not receive any assessment interview during the telephone screen.
  Participants randomized to this arm will receive the 8-week internet-delivered cognitive behaviour therapy (ICBT) course for alcohol misuse with guidance from a health educator through regular weekly online messages. Participants may also be contacted through emails and phone calls. The team of guides consists of registered social workers, psychologists, and graduate students, with experience delivering ICBT.
  Interventions: Behavioral: Guidance; Behavioral: ICBT for alcohol misuse
- ICBT for alcohol misuse: No Assessment Interview/No Guidance (Experimental): The client will not receive any assessment interview during the telephone screen.
  Participants randomized to this arm will receive the 8-week internet-delivered cognitive behaviour therapy (ICBT) course for alcohol misuse. Participants are able to contact the Online Therapy Unit regarding any technical issues with logging onto the site. However, no guidance from a health educator will be provided. Clients will be monitored by providing brief measures on alcohol and depression each week. However, clients will only be contacted if there is a significant clinical issue requiring attention (e.g., sudden increase in symptoms of depression and suicidal ideation).
  Interventions: Behavioral: ICBT for alcohol misuse

INTERVENTIONS:
Behavioral: Assessment Interview — An interviewer will administer a pre-treatment assessment interview. This 30-45 minute interview will be performed after randomization immediately after the initial telephone screen, where the interviewer will use the AUD section of the SCID-5.
  Arms: ICBT for alcohol misuse: Assessment Interview/Guidance; ICBT for alcohol misuse: Assessment Interview/No Guidance
Behavioral: Guidance — Guidance from a health educator through regular weekly online messages. Participants may also be contacted through emails and phone calls. The team of guides consists of registered social workers, psychologists, and graduate students, with experience delivering ICBT.
  Arms: ICBT alcohol misuse: No Assessment Interview/Guidance; ICBT for alcohol misuse: Assessment Interview/Guidance
Behavioral: ICBT for alcohol misuse — The 8-week internet-delivered cognitive behaviour therapy (ICBT) course for alcohol misuse. The course consists of 12 lessons distributed across 8 weeks (1 to 2 lessons a week).

SUMMARY:
Internet-delivered cognitive behaviour therapy (ICBT) shows considerable promise as a convenient treatment for alcohol misuse. ICBT may differ in whether the user works alone (self-guided) or along with an individual who guides treatment (e.g., therapist/health educator). Guided ICBT involves completing online lessons over several weeks coupled with support from a guide in the form of emails, online messages and/or brief telephone calls. Self-guided ICBT allows users to complete lessons by themselves without any contact with a guide. In some studies, guided-ICBT has shown greater reductions in alcohol consumption than self-guided ICBT. Further, some research on alcohol treatment shows that assessment in itself may have an effect on alcohol consumption, a phenomenon referred to in the literature as "assessment reactivity". It is believed that verbalizing one's drinking problems to another person might lead to greater realization of the problem extent and severity, which in turn can lead to initiation of the change process. Experimental studies have shown that extended and frequent assessments lead to greater alcohol reductions compared to brief and infrequent assessments.

Although ICBT for alcohol misuse is an attractive treatment option, it is not often available to clients as part of routine care. The Online Therapy Unit at the University of Regina is currently exploring extending services to include guided ICBT for alcohol misuse. The Unit has been providing treatment in ICBT for depression and anxiety as well as various health conditions since 2010 and has offered treatment to ~4200 individuals. The purpose of this study is to evaluate ICBT for individuals with alcohol misuse within the routine online clinic, and to investigate ways to optimize future modes of delivery. Of specific interest in this study, is how outcomes vary depending on whether or not weekly guidance from a health educator is available and whether or not an initial extended assessment telephone call is included or not compared to a briefer screening telephone call. Of interest will also be if the extended assessment leads to greater alcohol reductions and higher motivation pre-treatment.

DETAILED DESCRIPTION:
Alcohol misuse refers to alcohol consumption that causes harm to the drinker, others, and/or greater society. Internet-delivered cognitive behaviour therapy (ICBT) shows considerable promise as a convenient treatment for alcohol misuse. The overall goal of ICBT for alcohol misuse is typically behavioural change measured in terms of reduction of drinks consumed, as opposed to abstinence. The design of these interventions may differ in whether the user works alone (self-guided) or along with an individual who guides treatment (e.g., therapist/health educator). Guided ICBT involves completing online lessons over several weeks coupled with support from a guide in the form of emails, online messages or brief telephone calls. Self-guided ICBT allows users to complete lessons by themselves without any contact with a guide. In some studies, guided-ICBT has shown greater reductions in alcohol consumption than self-guided ICBT. Further, some research on alcohol treatment shows that assessment in itself may have an effect on alcohol consumption, a phenomenon referred to in the literature as "assessment reactivity". It is believed that verbalizing one's drinking problems to another person might lead to greater realization of the problem extent and severity, which in turn can lead to initiation of the change process. Experimental studies have shown that extended and frequent assessments lead to greater alcohol reductions compared to brief and infrequent assessments.

Although ICBT for alcohol misuse is an attractive treatment option, it is not often available to clients as part of routine care. The Online Therapy Unit at the University of Regina is currently exploring extending services to include guided ICBT for alcohol misuse. The Unit has been providing treatment in ICBT for depression and anxiety as well as various health conditions since 2010 and has offered treatment to ~4200 individuals. The purpose of this study is to evaluate ICBT for individuals with alcohol misuse, and to investigate ways to optimize future modes of delivery. Of specific interest in this study, is how outcomes vary depending on whether or not weekly guidance from a health educator is available and whether or not an initial extended assessment telephone call is included or not compared to a briefer screening telephone call.

Clients will be recruited online, through use of Google Ads and/or Facebook ads. Clients may also learn of the course from providers/organizations who will be informed of the study through posters, emails, and phone calls. All interested clients will be directed to the study website (www.onlinetherapyuser.ca) to complete an online screening questionnaire. As part of this questionnaire, they will be presented with a consent form explaining the screening protocol. After consent is given, clients will be assessed for eligibility using an online screening questionnaire. The online screening questionnaire captures demographic information (e.g., sex, ethnicity, location), contact details (e.g., telephone number, email address), information about alcohol, depression and other mental health issues, and background information needed to deliver therapy (e.g., medical history, mental health history, symptoms).

Once clients have been assessed for eligibility through the online screening questionnaire, they will be asked to book a telephone interview with unit staff. During the telephone screening interview, clients will be asked a series of follow-up questions to the online screening questionnaire to ensure eligibility as per exclusion criteria. Clients who meet any of the exclusion criteria during the online telephone screening interview will be referred to more appropriate mental health services. Clients who are excluded in the screening questionnaire by reporting a low score on either TLFB or AUDIT, or a high score on PHQ-9, will be informed about relevant treatment options and will be offered unguided ICBT with no assessment interview. Clients who are included in the study, will be randomized by the interviewer, while the client is still on the phone, to one of four conditions. The two factors in the trial are:

Factor 1: Guidance (yes or no)

Factor 2: Assessment interview (yes or no)

As this is a factorial trial with two factors, each client will be randomized to one of four conditions:

Condition 1: Assessment interview and Guidance Condition 2: Assessment Interview and No Guidance Condition 3: No Assessment Interview and Guidance Condition 4: No Assessment Interview and No Guidance

After the randomization those randomized to either condition that includes assessment interview will receive this interview immediately. The assessment interview consists of the Alcohol Use Disorder section of Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders 5 (SCID5). Clients will then be provided a user-name and temporary password, Those randomized to conditions with no assessment interview will be provided user-name and password immediately after the randomization.

All clients will have access to the ICBT course on the second Monday after the screening interview, regardless of whether they have been randomized to assessment interview or not.

Before accessing the ICBT course with user-name and password, clients will be presented with a consent form that explains the nature of treatment, as well as a pre-treatment questionnaire, where participants will complete questions about alcohol consumption in the preceding week, depression and motivation to change.

All clients will receive the Alcohol Change Course, an internet intervention targeting alcohol misuse. The course is an adaptation of a program originally developed in Switzerland. The program has been adapted to better fit the programs that are commonly used at the Online Therapy Unit (8 weeks in length, gradual time release, downloadable exercises, wide range in age). Patient partners have also studied the program and provided feedback, which has led to additional changes. It comprises 12 online lessons (1 to 2 lessons per week over 8 weeks), and the content is based on cognitive behaviour therapy and relapse prevention. Materials are presented in a didactic (i.e., text-based with visual images) and case-enhanced learning format (i.e., educational stories demonstrate the application of skills). All clients are presented with worksheets at the end of each lesson that contain exercises that facilitate skill acquisition. In all conditions, lessons will be released gradually in a standardized order over 8 weeks with regular automatic emails informing clients about upcoming lessons. Clients will complete outcome questionnaires at screening, baseline (pre-treatment), 8 weeks (post-treatment) and at 3, 6 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Timeline Followback (TLFB; preceding week alcohol consumption) > 13 drinks
* Alcohol Use Disorders Identification Test (AUDIT) > 7

Exclusion Criteria:

* Severe depression (measured by scoring > 23 on PHQ-9)
* Suicidal ideation (measured by scoring > 2 to question 9 of PHQ-9)
* Severe mental health or medical conditions
* Severe drug use problems (measured by scoring > 24 on Drug Use Disorders Identification Test [DUDIT] or clinical assessment)
* Low motivation to do, or concerns regarding, online treatment
* Ongoing or impending significant mental health treatment
* Not residing in Canada for the duration of treatment
* Lack of or inconsistent access to a computer and internet at home or private place for the duration of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Drinks preceding week as measured by Timeline Followback (TLFB) | Screening, Pre-treatment, 4 weeks (mid-treatment), 8 weeks (post-treatment), 3 months after treatment, 6 months after treatment, 12 months after treatment
  Change in preceding week alcohol consumption in terms of the total number of standard drinks consumed on each day during the previous 7 days.
Heavy drinking days preceding week as measured by Timeline Followback (TLFB). | Screening, Pre-treatment, 4 weeks (mid-treatment), 8 weeks (post-treatment), 3 months after treatment, 6 months after treatment, 12 months after treatment
  Change in preceding week alcohol consumption in terms of the total number of heavy drinking days during the previous 7 days.

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT). | Screening, 8 weeks (post-treatment), 3 months after treatment, 6 months after treatment, 12 months after treatment
  Change in alcohol-related problems and behaviours measured by total AUDIT score which can range from 0 to 40. Greater score indicates greater alcohol problems (worse outcome)
Penn Alcohol Craving Scale | Screening, 8 weeks (post-treatment), 3 months after treatment, 6 months after treatment, 12 months after treatment
  Change in alcohol craving as measured by a total score ranging between 0 to 30. Higher scores indicate greater craving (worse outcome).
Brief Situational Confidence Questionnaire (BSCQ). | Screening, 8 weeks (post-treatment), 3 months after treatment, 6 months after treatment, 12 months after treatment
  Change in confidence in resisting drinking urges in 8 situations rated from 0 to 100, rendering a sum score of 0-800. Higher scores indicate greater confidence (better outcome). There are 8 subscales, one for each item, assessed on a scale of 0-100. Thus, each subscale has a sum score of 0-100-. A higher score indicates greater confidence on the subscale.
Generalized Anxiety Disorder 7-item (GAD-7) | Screening, 8 weeks (post-treatment), 3 months after treatment, 6 months after treatment, 12 months after treatment
  Change in total GAD-7 anxiety score which can range from 0 to 21. Higher scores indicate greater anxiety (worse outcome)
Patient Health Questionnaire (PHQ-9) | Screening (Pre-treatment), 4 weeks (mid-treatment), 8 weeks (post-treatment), 3 months after treatment, 6 months after treatment, 12 months after treatment
  Change in total PHQ-9 score which can range from 0 to 27. Higher scores indicate greater depression (worse outcome)
Sheehan Disability Scale | Screening, 8 weeks (post-treatment), 3 months after treatment, 6 months after treatment, 12 months after treatment
  Change in three scores assessing functional impairment in three domains: 1) work/school, 2) social and 3) family life (each domain score ranges from 0 to 10, rendering a sum score of 0-30). Higher score indicates greater ability on the specified domain score (better outcome). Each domain score (subscale) renders a sum score of 0-10.
Treatment Credibility and Expectancy Scale | 4 weeks (mid-treatment)
  Measures the participant's thoughts and feelings about the treatment and the treatment's effectiveness in reducing participant's symptoms and increasing participant's functioning. Consists of 6 items. The first three of these and the 5th render a score of 1- 9. The other three questions render a score of 0-10. There are two subscales; 1) treatment credibility and 2) treatment expectancy. The first three questions are summed to render a score on the credibility subscale (0-27). The last three questions, the expectancy subscale, render a score of 0-29.
Readiness to Change Questionnaire Treatment Version (RCQ-TV) | Screening (Pre-treatment)
  Measures participants' motivation to change their drinking behaviours and determines at which stage of the Stages of Change model they are in (precontemplation, contemplation, or action). There is no sum score. Instead the items related to each stage are summed, and the individual is allocated to the stage that has the greatest score out of these three. (For more information about the scoring of this instrument, see Heather & Hönekopp, 2009).
Evaluation and Negative Effects Questionnaire | 8 weeks (post-treatment)
  Measures negative effects experienced by participants during treatment. This questionnaire has been developed by the research team, and does not have a sum score.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sundstrom C, Peynenburg V, Chadwick C, Thiessen D, Wilhems A, Nugent M, Keough MT, Schaub MP, Hadjistavropoulos HD. Optimizing internet-delivered cognitive behaviour therapy for alcohol misuse-a randomized factorial trial examining effects of a pre-treatment assessment interview and guidance. Addict Sci Clin Pract. 2022 Jul 23;17(1):37. doi: 10.1186/s13722-022-00319-0. PMID 35871010
- [Derived] Sundstrom C, Hadjistavropoulos H, Wilhelms A, Keough M, Schaub M. Optimizing internet-delivered cognitive behaviour therapy for alcohol misuse: a study protocol for a randomized factorial trial examining the effects of a pre-treatment assessment interview and health educator guidance. BMC Psychiatry. 2020 Mar 17;20(1):126. doi: 10.1186/s12888-020-02506-2. PMID 32183769